CLINICAL TRIAL: NCT00151723
Title: Subclinical Hyperthyroidism "To Treat or Not to Treat?" A Dutch Multicenter Trial
Brief Title: Does Radioiodine Treatment Prevent Atrial Fibrillation and Bone Loss in Endogenous Subclinical Hyperthyroidism?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SUBstudie
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2007-07-18 (Estimated); Status verified 2005-09

CONDITIONS: Hyperthyroidism
Keywords: endogenous subclinical hyperthyroidism
MeSH Terms: conditions — Hyperthyroidism | interventions — Therapeutics

INTERVENTIONS:
Procedure: treatment with 131I

SUMMARY:
Subclinical hyperthyroidism is defined as the presence of serum free thyroxine (T4) and triiodothyronine (T3) levels within the reference range and a reduced serum thyrotrophin (TSH) level. Evidence is accumulating that it has important clinical effects. The SUBstudy is a randomised, Dutch multicenter trial to study whether radioiodine treatment prevents the development of atrial fibrillation and prevents decreases in bone mineral density in patients with endogenous subclinical hyperthyroidism.

ELIGIBILITY:
Inclusion Criteria:

* Subclinical hyperthyroidism [TSH ≤ 0.1 mU/L, fT4 and T3 within the normal range of the own laboratory (determined 2 times in own laboratory) with an interval of at least 2 months].
* Endogenous cause of subclinical hyperthyroidism limited to autonomous adenoma or multinodular goiter (diagnosis made by the attending physician, based on palpation and the result of a thyroid scintigram).
* Informed consent.

Exclusion Criteria:

* Medication with anti-thyroid drugs in the last 3 months (also not allowed during follow-up); thyroid hormone in the last 3 months (allowed during follow-up, but TSH levels should be kept between 0.1 mU/L and the upper limit of normal in the own laboratory); and oral glucocorticoids in the last 3 months (allowed during follow-up when absolutely necessary, but patients in whom glucocorticoids are started cannot be evaluated with respect to changes in bone mineral density [BMD]).
* Radioiodine therapy in the past.
* Iodine-induced subclinical hyperthyroidism.
* Pituitary or hypothalamic insufficiency.
* Pregnancy.
* Age <= 40 years.
* Severe non-thyroidal illness.
* Drug abuse.
* Unstable angina pectoris, (history of) atrial fibrillation, (history of) congestive heart failure.
* (History of) osteoporotic fracture(s).
* Patients younger than 70 years of age with a bone mineral density T-score < - 2.5 standard deviations (SD), or older than 70 years of age with a bone mineral density Z-score < 1.0 SD. (These patients can be randomized but in case it is decided to treat them with anti-osteoporotic drugs they cannot be evaluated with respect to changes in BMD.)
* Use of betablockers in the last three months. (These patients can be randomised but cannot be evaluated with respect to general and cardiac symptoms. The same applies to patients in whom betablockers are started during follow up.)
* Other symptoms or signs of hyperthyroidism or obstruction of vital structures which, in the opinion of the attending physician, require active treatment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-04

PRIMARY OUTCOMES:
To provide evidence that restoration of euthyroidism (normal TSH) improves thyrotoxic symptoms and signs and quality of life and lowers the risk of subsequent atrial fibrillation and bone loss in subjects with endogenous subclinical hyperthyroidism

CONTACTS AND LOCATIONS:
Overall Officials: Ad Hermus, MD, Prof, Principal Investigator — Radboud University Medical Center
Locations (5):
- Netherlands (5):
  - Academical Medical Centre Amsterdam, Amsterdam
  - Martini Ziekenhuis Groningen, Groningen
  - University Hospital Groningen, Groningen
  - Radboud University Medical Centre Nijmegen, Nijmegen
  - Maxima Medisch Centrum, Veldhoven

REFERENCES:
- [Background] Hoogendoorn EH, Wiersinga WM, Prummel MF, den Heijer M, Corstens FH, Hermus AR. [Subclinical hypothyroidism; the start of a clinical trial into the usefulness of treatment with radioactive iodine]. Ned Tijdschr Geneeskd. 2004 May 8;148(19):953-4. Dutch. PMID 15160563